CLINICAL TRIAL: NCT05686447
Title: Screening and Therapeutic Monitoring of Multiple Myeloma by MALDI-TOF MS Analysis
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Hongwei Zhou, Professor, Zhujiang Hospital
Other Study IDs: Zhujianghjd
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Monoclonal Gammopathies; Multiple Myeloma; M-protein
Keywords: M-protein
MeSH Terms: conditions — Paraproteinemias; Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple myeloma: Multiple myeloma (MM) is a hematologic malignant tumor characterized by abnormally cloned plasma cells in bone marrow, whose growth can lead to destructive bone injury, acute kidney injury, anemia, and hypercalcemia.
  Interventions: Other: Observational studies, no intervention
- Healthy control: Individuals in good health without obvious disease and with normal physical examination report; Avoid people who have not suffered from major chronic diseases in recent years, such as hypertension, diabetes, chronic kidney disease, etc; controls were appropriately selected that matched cases for age and sex.
  Interventions: Other: Observational studies, no intervention

INTERVENTIONS:
Other: Observational studies, no intervention — Observational studies, no intervention

SUMMARY:
To provide a comprehensive MALDI-TOF mass spectrometry method for detecting, characterizing, and quantifying M-protein, and to track M-protein in a very sensitive and specific manner during patient treatment, providing a more precise test for diagnosing disease and monitoring patient response to treatment.

DETAILED DESCRIPTION:
M-protein is a serum biomarker directly related to clonal plasma cell load in Multiple myeloma (MM) patients and can be used as a diagnostic marker to make out disease and a quantitative marker to track disease progression and response to treatment. Identification, typing and quantification of M-proteins are useful for initial diagnosis of disease, risk stratification and monitoring of response to treatment. Although the determination of M-protein can be used as an auxiliary diagnosis of multiple myeloma, the early diagnosis and risk assessment of MM still lack convenient and effective tools for large-scale screening. In recent years, the use of matter-assisted laser desorption/ionization time-of-flight mass spectrometry (MALDI-TOF MS) for proteomic analysis of complex biological mixtures has attracted extensive attention, and has become one of the most promising methods for the detection of m proteins. In this study, we screened the population by MALDI mass spectrometry in order to detect low level circulating M-protein by a faster and more sensitive method.

ELIGIBILITY:
Inclusion Criteria:(1) Inclusion criteria for cases: Serum samples from related people diagnosed with multiple myeloma were included in MALDI-TOF-MS analysis by serum protein electrophoresis (SPEP), serum immunofixation electrophoresis (IFE), Ig isotype detection and other methods. (2) Inclusion criteria of the controls were as follows: individuals in good health without obvious disease and with normal physical examination report; Avoid people who have not suffered from major chronic diseases in recent years, such as hypertension, diabetes, chronic kidney disease, etc; controls were appropriately selected that matched cases for age and sex.

-

Exclusion Criteria: samples with incomplete sample information and untraceable source; Samples whose sample volume is insufficient for testing; Samples that do not meet the requirements for sample collection and storage

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All the patients with Multiple myeloma hospitalized in Zhujiang hospital will be eligible to be enrolled. Also, their age- and sex- matched healthy controls making a physical examination in Zhujiang hospital will be eligible to be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
M-protein | baseline
  M-protein in urine and serum detected using MALDI-TOF Mass Spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Zhou, Professor, Study Chair — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No